CLINICAL TRIAL: NCT03391011
Title: Non-contact Intraoperative Optical Imaging During Neurosurgical Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Victor Yang, Senior Scientist, Physical Sciences Platform, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 086-2015
Record Dates: First submitted 2017-12-18; First posted 2018-01-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Computer-assisted Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBL Experimental Navigation System (Experimental): As this is a single arm trial, all participants receive treatment.
  Interventions: Device: BBL Experimental Navigation System

INTERVENTIONS:
Device: BBL Experimental Navigation System — Comparison of accuracy of screw placement using experimental system while monitored by clinically approved system.

SUMMARY:
For a significant number of patients suffering from back pain, even basic daily activities become impossible. It is at this time that spinal surgery becomes necessary in order to improve the patient's quality of life. To combat these symptoms, surgical implants (e.g. pedicle screws, rods, etc.) are used to aid in stabilizing and correcting the deformities of the spine, particularly after spinal decompression. The clinical need for spinal surgery is compounded by current and continuing demographic trends. As the general population continues to age, the number of orthopaedic surgical interventions is expected to rise drastically. Therefore, a significant opportunity exists for the implementation of surgical guidance technologies, for orthopaedic procedures, to combat this overwhelming health care burden.

DETAILED DESCRIPTION:
The hypothesis is that optical visualization of surgically exposed anatomy with the Biophotonics and Bioengineering Lab (BBL) surgical navigation prototype, when registered with pre-operative imaging (CT or MRI), can accurately estimate subsurface anatomy and allow tracking the position of surgical instruments in real-time, using an intraoperative non-contact optical imaging system during spinal surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age, able to provide consent, or has substitute decision maker available to consent.
* Scheduled to undergo spinal instrumentation surgery involving pedicle or lateral mass screw insertion.
* Scheduled for pre-operative CT scan and the surgical plan includes open exposure of the posterior bony elements of two or more level(s) of the vertebra(e).
* No contra-indication for a post-operative CT scan.

Exclusion Criteria:

* Previous spinal decompression with significant laminectomy performed at the level intended for instrumentation.
* Previous spinal instrumentation with significant metallic artefact on pre-operative CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03-13 (Actual); Primary Completion 2019-03-13 (Estimated); Study Completion 2019-03-13 (Estimated)

PRIMARY OUTCOMES:
Pilot hole and screw trajectory accuracy as compared between post-operative CT and intraoperative images | Within 1 week of screw placement
  Comparison and quantification of accuracy of pilot holes including entry point and trajectory as taken from experimental navigation system as compared to absolute (or actual) entry point and trajectory of screws as determined by post-operative computed tomography scans.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yee, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre; Victor XD Yang, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merloz P, Tonetti J, Eld A, et al, Computer-assisted versus manual spine surgery: Clinical report, Springer Berlin, 1997.
- [Background] Rampersaud YR, Simon DA, Foley KT. Accuracy requirements for image-guided spinal pedicle screw placement. Spine (Phila Pa 1976). 2001 Feb 15;26(4):352-9. doi: 10.1097/00007632-200102150-00010. PMID 11224881
- [Background] Zdichaversusky M, Blauth M, Knop C, Graessner M, Herrmann H, Krettek C, Bastian L, Accuracy of Pedicle Screw Placement in Thoracic Spine Fractures, European Journal of Trauma, 30:234-240, 2004
- [Background] Waters JD, Gonda DD, Reddy H, Kasper EM, Warnke PC, Chen CC. Diagnostic yield of stereotactic needle-biopsies of sub-cubic centimeter intracranial lesions. Surg Neurol Int. 2013 Apr 17;4(Suppl 3):S176-81. doi: 10.4103/2152-7806.110677. Print 2013. PMID 23682345
- [Background] Labadie RF, Davis BM, Fitzpatrick JM. Image-guided surgery: what is the accuracy? Curr Opin Otolaryngol Head Neck Surg. 2005 Feb;13(1):27-31. doi: 10.1097/00020840-200502000-00008. PMID 15654212
- [Background] Snyderman C, Zimmer LA, Kassam A. Sources of registration error with image guidance systems during endoscopic anterior cranial base surgery. Otolaryngol Head Neck Surg. 2004 Sep;131(3):145-9. doi: 10.1016/j.otohns.2004.03.002. PMID 15365528
- [Background] Pillai P, Sammet S, Ammirati M. Application accuracy of computed tomography-based, image-guided navigation of temporal bone. Neurosurgery. 2008 Oct;63(4 Suppl 2):326-32; discussion 332-3. doi: 10.1227/01.NEU.0000316429.19314.67. PMID 18981839
- [Background] Mathew JE, Mok K, Goulet B. Pedicle violation and Navigational errors in pedicle screw insertion using the intraoperative O-arm: A preliminary report. Int J Spine Surg. 2013 Dec 1;7:e88-94. doi: 10.1016/j.ijsp.2013.06.002. eCollection 2013. PMID 25694911
- [Background] Rajasekaran S, Vidyadhara S, Ramesh P, Shetty AP. Randomized clinical study to compare the accuracy of navigated and non-navigated thoracic pedicle screws in deformity correction surgeries. Spine (Phila Pa 1976). 2007 Jan 15;32(2):E56-64. doi: 10.1097/01.brs.0000252094.64857.ab. PMID 17224800